CLINICAL TRIAL: NCT06059131
Title: Randomized Controlled and Double-blinded Study of the Effect of a Specific Aquaporin-1 Inhibitor, Bacopaside II (KeenMind®), on Vascular Oxidative Stress in Healthy Volunteers
Brief Title: Effect of a Specific Aquaporin-1 Inhibitor on Vascular Oxidative Stress in Healthy Volunteers
Acronym: Bacoxy_II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2023/11JAN/014
Record Dates: First submitted 2023-08-01; First posted 2023-09-28 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Oxidative Stress; Cardiovascular Diseases; Bacopaside II; Bacopa Monnieri; Endothelial Dysfunction; Aquaporin 1; AQP1
Keywords: vascular oxidative stress; aquaporin 1; AQP1; peroxiporin; H2O2; hydrogen peroxide; cardiovascular diseases; Bacopa monnieri; Bacopaside II; endothelial dysfunction
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: 2 arms : placebo vs verum
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization is performed by an independent statistical service. The randomization list will be transferred to the hospital pharmacy. The pharmacists will be responsible for the delivery of the capsules (placebo vs. verum). Neither the investigator nor the participant will be aware of the treatment. The code will be unmasked at the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KeenMind (Experimental)
  Interventions: Other: KeenMind
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: KeenMind — 320 mg/d (2 capsules/d) during 3 months
  Other Names: Bacopa monnieri
  Arms: KeenMind
Other: Placebo — 320 mg/d (2 capsules/d) during 3 months
  Arms: Placebo

SUMMARY:
Bacoxy_II study aims to evaluate the efficacy of a standardized Bacopa monnieri extract, KeenMind®, on vascular oxidative stress.

DETAILED DESCRIPTION:
The food supplement Bacopa monnieri is a plant used in Ayuverda medicine, especially in the treatment of chronic neurological disease with cognitive impairment and memory disorders and for stress management.

Bacopa monnieri contains several Bacosides including Bacopaside II, a specific inhibitor of aquaporin 1 (AQP1), the main water chanel found in mammalian cardiovacular tissues.

AQP1, more than a water chanel, is a peroxiporin able to facilitate the passage of H2O2.

AQP1 is present in myocyte, endothelial and red blood cells. Concerning the endothelial function, analyses in the FATH laboratory (IREC - UCLouvain), confirm the attenuation of H2O2 transport by AQP1 through Bacopaside II in red blood cells but also in endothelial cells.

As H2O2 is involved in oxidative stress mechanisms and endothelial dysfunction, the investigators hypothezised that the oral intake of Bacopa monnieri containing the Bacopaside II could induce an inhibition of AQP1 and attenuate the passage of H2O2 leading to an attenuation of vascular oxidative stress and endothelial function.

In order to answer to this question, the investigators set up the Bacoxy_II clinical study, that is a double-blind, prospective, interventional and controlled study. The study will last 4 months, including 3 months of treatment and 1 month of post-treatment follow-up. This study will include 2 groups of 20 volunteers: one group will receive a dose of 320 mg/d of Bacopa monnieri and the other group will receive the placebo treatment.

ELIGIBILITY:
Inclusion Criteria:

- healthy volunteers

Exclusion Criteria:

* any chronic disease
* use of chronic drugs or food supplements
* smoking

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Ex vivo DCFDA test on red blood cells (RBCs) | Baseline (V0), 3 months (V1), 4 months (V2)
  DCFA is a probe used to assess the presence of intracellular ROS. Red blood cells are incubated with DCFA and H2O2. In cells, DCFA is transformed into DCF in the presence of ROS such as H2O2 and the intensity of the emitted signal can be measured by FACS. This technique allows us to measure kinetically the entry of H2O2 by AQP1 in RBCs
Nitrosylated hemoglobin (HbNO) | Baseline (V0), 3 months (V1), 4 months (V2)
  Oxidative stress is involved in the decreased bioavailability of nitric oxide (NO). HbNO a complexe used to assess NO bioavailability. HbNO can be quantify by electron paramagnetic resonance spectroscopy.
Lipid peroxydes | Baseline (V0), 3 months (V1), 4 months (V2)
  Lipid peroxidation is oxidative damage that affects cellular membranes, lipoproteins, and other molecules that contain lipids in conditions with oxidative stress. Assessement of changes in lipid peroxides level during the study is a reflect of oxidative status. Lipid peroxydes are measured by an ELISA test.
EndoPAT | Baseline (V0), 3 months (V1), 4 months (V2)
  Endo-PAT is a non-invasive technique to assess peripheral arterial tone following a reactive hyperemia phenomenon. Using probes placed on the fingertips, EndoPAT measures changes in vascular tone mediated by the endothelium following reactive hyperemia induced by forearm occlusion using a cuff.

SECONDARY OUTCOMES:
C-reactive protein (CRP) | Baseline (V0), 3 months (V1), 4 months (V2)
  C-reactive protein is a marker of inflammation. unit: mg/L The CRP assesses the inflammatory state of an individual. CRP is measured in the serum after a blood sampling.
Blood count | Baseline (V0), 3 months (V1), 4 months (V2)
  The hemogram is a quantitative and qualitative analysis of blood constituents. This test is performed to reiterate the known safety of Bacopa monnieri on the systemic circulation after oral ingestion. The haemogram includes the following measurements: haemoglobin (g/L), haematocrit (g/L) and red blood cells (10^6/µL).
Ion count | Baseline (V0), 3 months (V1), 4 months (V2)
  As Bacopa monnieri has a diuretic effect, an ionic count will help assess the concentration of electrolytes in the blood. The ion count includes the following measurements: Sodium (mM), potassium (mM), chloride (mM), bicarbonate (mM).
Lipid count | Baseline (V0), 3 months (V1), 4 months (V2)
  To assess the effect of Bacopa monnieri on the lipid profile, we measure blood lipids. Lipids include total cholesterol (mg/dL), HDL cholesterol (mg/dL), LDL cholesterol (mg/dL) and triglycerides (mg/dL).
Liver function | Baseline (V0), 3 months (V1), 4 months (V2)
  Liver function will be assessed to verify the known safety of Bacopa monnieri. Liver function includes: transaminase level (U/L) and gamma-glutamyl-transferase level (U/L).
Kidney function | Baseline (V0), 3 months (V1), 4 months (V2)
  Renal function will be assessed to reiterate the known safety of Bacopa monnieri. Renal function includes the following measurements: creatinine (mg/dl), urea (mg/dl) and glomerular filtration rate (ml/min/m²).
HOMA index | Baseline (V0), 3 months (V1), 4 months (V2)
  The HOMA index will be used to assess changes in insulin sensitivity over the course of the study. The HOMA index is calculated as follows: Fasting blood glucose (mmol/L) * Fasting insulin (mui/mL)/22.5. To calculate this index, we measure fasting blood glucose (mg/dL) and fasting insulin (pmol/L). An index >2.4 is a diagnostic of insulin resistance.
Body mass index, fat mass, lean mass, | Baseline (V0), 3 months (V1), 4 months (V2)
  To assess changes in body composition over the course of the study, we will be using impedance measurement technology. Impedance analysis is used to calculate lean mass (%), fat mass (%) and fluid volume (%).
Waist and hip circumference ratio | Baseline (V0), 3 months (V1), 4 months (V2)
  To assess changes in body composition over the course of the study, we measure waist and hip circumferences. We measure these circumferences using a tape measure in centimetres.

CONTACTS AND LOCATIONS:
Overall Officials: Virginie Montiel, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint Luc, Brussels, Belgique, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pravina K, Ravindra KR, Goudar KS, Vinod DR, Joshua AJ, Wasim P, Venkateshwarlu K, Saxena VS, Amit A. Safety evaluation of BacoMind in healthy volunteers: a phase I study. Phytomedicine. 2007 May;14(5):301-8. doi: 10.1016/j.phymed.2007.03.010. Epub 2007 Apr 17. PMID 17442556
- [Background] Stough C, Downey LA, Lloyd J, Silber B, Redman S, Hutchison C, Wesnes K, Nathan PJ. Examining the nootropic effects of a special extract of Bacopa monniera on human cognitive functioning: 90 day double-blind placebo-controlled randomized trial. Phytother Res. 2008 Dec;22(12):1629-34. doi: 10.1002/ptr.2537. PMID 18683852
- [Background] Dave UP, Dingankar SR, Saxena VS, Joseph JA, Bethapudi B, Agarwal A, Kudiganti V. An open-label study to elucidate the effects of standardized Bacopa monnieri extract in the management of symptoms of attention-deficit hyperactivity disorder in children. Adv Mind Body Med. 2014 Spring;28(2):10-5. PMID 24682000
- [Background] Montiel V, Leon Gomez E, Bouzin C, Esfahani H, Romero Perez M, Lobysheva I, Devuyst O, Dessy C, Balligand JL. Genetic deletion of aquaporin-1 results in microcardia and low blood pressure in mouse with intact nitric oxide-dependent relaxation, but enhanced prostanoids-dependent relaxation. Pflugers Arch. 2014 Feb;466(2):237-51. doi: 10.1007/s00424-013-1325-x. Epub 2013 Jul 20. PMID 23873354
- [Background] Montiel V, Bella R, Michel LYM, Esfahani H, De Mulder D, Robinson EL, Deglasse JP, Tiburcy M, Chow PH, Jonas JC, Gilon P, Steinhorn B, Michel T, Beauloye C, Bertrand L, Farah C, Dei Zotti F, Debaix H, Bouzin C, Brusa D, Horman S, Vanoverschelde JL, Bergmann O, Gilis D, Rooman M, Ghigo A, Geninatti-Crich S, Yool A, Zimmermann WH, Roderick HL, Devuyst O, Balligand JL. Inhibition of aquaporin-1 prevents myocardial remodeling by blocking the transmembrane transport of hydrogen peroxide. Sci Transl Med. 2020 Oct 7;12(564):eaay2176. doi: 10.1126/scitranslmed.aay2176. PMID 33028705